CLINICAL TRIAL: NCT04412876
Title: Comparisons of the Impact of Duloxetine Versus Imipramine on Therapeutic Efficacy, Psychological Distress, Sexual Function, Urethral and Bladder Wall Structure and Blood Flow in Women With Stress Urinary Incontinence: a Randomized Controlled Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Failed to pass the Ministry of Science and Technology.
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109017-F
Record Dates: First submitted 2020-05-31; First posted 2020-06-02 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2021-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride; Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Experimental): Receive Duloxetine 30 mg treatment per day
  Interventions: Drug: Duloxetine
- Imipramine (Active Comparator): Receive Imipramine 25 mg treatment per day
  Interventions: Drug: Imipramine

INTERVENTIONS:
Drug: Duloxetine — Duloxetine 30 mg qd
  Arms: Duloxetine
Drug: Imipramine — Imipramine 25mg qd
  Arms: Imipramine

SUMMARY:
To assess the impact of Duloxetine and Imipramine on therapeutic efficacy, psychological distress, sexual function, bladder wall structure and blood flow in women

DETAILED DESCRIPTION:
To assess the impact of Duloxetine and Imipramine on therapeutic efficacy, psychological distress, sexual function, bladder wall structure and blood flow in women

ELIGIBILITY:
Inclusion Criteria:

- Stress urinary incontinence

Exclusion Criteria:

1. Take monoamine oxidase
2. Myocardial infarction critical,cardiovascular insufficiency (such as room blocking, arrhythmia, blood-soaked heart failure, myocardial infarction, stroke and excessive heartbeat).
3. Allergy to duloxetine or imipramine
4. Uncontrolled angular glaucoma patients
5. Pregnant women

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
the score of International Consultation on Incontinence Questionnaire-Urinary Incontinence | 8 weeks
  Between-group difference in the score of International Consultation on Incontinence Questionnaire-Urinary Incontinence

SECONDARY OUTCOMES:
the score of Urgency Severity Scale | 8 weeks
  Between-group difference in the score of Urgency Severity Scale

OTHER OUTCOMES:
the score of Overactive Bladder Symptom Score | 8 weeks
  Between-group difference in the score of Overactive Bladder Symptom Score
the score of King's health questionnaires | 8 weeks
  Between-group difference in the score of King's health questionnaires
the score of Brief symptom rating scale | 8 weeks
  Between-group difference in the score of Brief symptom rating scale
the score of Female sexual function index | 8 weeks
  Between-group difference in the score of Female sexual function index
Blood flow index of the bladder | 8 weeks
  Between-group difference in the changes of blood flow index of the bladder
Bladder wall thickness | 8 weeks
  Between-group difference in the changes of Bladder wall thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No